CLINICAL TRIAL: NCT05857007
Title: CGM Utilization With IV Insulin EndoTool and Subcutaneous Insulin in the Neuro ICU
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00087771
Record Dates: First submitted 2023-04-27; First posted 2023-05-12 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus; Hyperglycemia
Keywords: CGM; IV insulin; EndoTool; subcutaneous insulin; continuous glucose monitoring; NeuroICU; critical care settings; Libre2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Libre 2.0 CGM in patients taking EndoTool IV insulin: Ten patients with Hyperglycemia or/and Diabetes in the neuro ICU requires IV insulin through EndoTool algorithm will wear Libre 2.0 CGM for either 14 days or their stay in the neuro ICU
  Interventions: Device: Libre 2.0 CGM in patients taking subcutaneous insulin with concomitant high dose glucocorticoids

INTERVENTIONS:
Device: Libre 2.0 CGM in patients taking subcutaneous insulin with concomitant high dose glucocorticoids — Ten patients with hyperglycemia or/and diabetes in the neuro ICU requires subcutaneous insulin with concomitant high dose glucocorticoids will wear Libre 2.0 CGM for either 14 days or their stay in the neuro ICU

SUMMARY:
The goal of this study (CGM utilization with IV Insulin EndoTool and Subcutaneous Insulin in the Neuro ICU) is to understand how CGM technology utilized in conjunction with EndoTool IV insulin could improve glycemic management in the NeuroICU, specifically in predicting and preventing hypoglycemic and hyperglycemic episodes with resultant improvement in patient morbidity and mortality. The second arm of the study will focus on how CGM technology utilized in patients on basal bolus subcutaneous insulin while on high dose glucocorticoids could impact glycemic management. The main questions it aims to answer are:

1. Is CGM technology data accurate compared to the current standard point of care among NeuroICU patients?
2. How CGM technology could improve glycemic management in the critical care setting, specifically in predicting and preventing hypoglycemic episodes with IV or subcutaneous insulin?
3. How CGM technology could help treating hyperglycemia in the NeuroICU with resultant improvement in patient morbidity, mortality, and length of stay?

DETAILED DESCRIPTION:
The study is comparing current standard of care blood glucose fingersticks or serum blood glucose collection to CGM data utilizing the Freestyle Libre 2.0 CGM. A recently conducted study of 8 critically ill patients with diabetes that wore Freestyle Libre 2.0 CGM's during their ICU stay demonstrated high test-retest reliability and acceptable accuracy when compared with arterial blood glucose measurements. The study aims to evaluate utilization of CGM technology and EndoTool in the critical care setting by recruiting a cohort of 10 participants with hyperglycemia and/or diabetes mellitus who are anticipated to require blood glucose monitoring and IV insulin to achieve adequate glycemic control while in the Neuro ICU. The study also aims to evaluate utilization of CGM technology and subcutaneous insulin by recruiting a cohort of 10 patients with a history of diabetes mellitus on high dose steroids who are anticipated to require blood glucose monitoring and treatment with basal bolus insulin.

Participants will be enrolled on admission to the Neuro ICU and have the CGM device placed. The study aims to evaluate CGM technology by comparison of glucose values obtained from the CGM to the serum or fingerstick blood glucose levels while the patient is either receiving IV insulin via EndoTool or subcutaneous insulin while on high dose glucocorticoids. Current standard of care with monitoring glycemic data utilizing point of care blood glucose fingersticks and serum glucose will be utilized for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Participants that are 18 years of age or older with hyperglycemia and/or diabetes mellitus with need of IV insulin management or subcutaneous insulin with concomitant high dose glucocorticoids who are admitted to the Neuro ICU at Atrium Health Wake Forest Baptist Hospital.

Exclusion Criteria:

* Pregnant women will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hyperglycemia and/or diabetes mellitus with need of IV insulin management or subcutaneous insulin with concomitant high dose glucocorticoids who are admitted to the Neuro ICU at Atrium Health Wake Forest Baptist Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of CGM technology- Neuro ICU patients with hyperglycemia, DKA or HHS and require IV insulin using the EndoTool software, will wear the freestyle Libre 2.0 CGM for either 14 consecutive days or their Neuro ICU admission. | Participants will wear CGM for either 14 consecutive days or duration of their Neuro ICU admission
  Neuro ICU patients with hyperglycemia, DKA or HHS and require IV insulin using the EndoTool software, will wear the freestyle Libre 2.0 CGM for either 14 consecutive days or their Neuro ICU admission. CGM data will be available in real time to monitor glucose during their hospitalization and studying if this data could improve insulin titration using the EndoTool software. Dosing of insulin will be performed utilizing standard of care fingerstick blood glucose values and not CGM data.
Feasibility of CGM technology in the critical care setting - monitor glucose during their hospitalization and studying if this data could improve subcutaneous insulin titration | Participants will wear CGM for either 14 consecutive days or duration of their Neuro ICU admission
  Neuro ICU patients with hyperglycemia, DKA or HHS and require subcutaneous insulin with concurrent high dose glucocorticoids, will wear the freestyle Libre 2.0 CGM for either 14 consecutive days or their Neuro ICU admission. CGM data will be available in real time to monitor glucose during their hospitalization and studying if this data could improve subcutaneous insulin titration . Dosing of insulin will be performed utilizing standard of care fingerstick blood glucose values and not CGM data.
Comparison of CGM with fingerstick blood glucose values in critical care setting. | Participants will wear CGM for either 14 consecutive days or duration of their Neuro ICU admission
  Neuro ICU patients with hyperglycemia, DKA or HHS and require either EndoTool IV insulin or subcutaneous insulin with concurrent high dose glucocorticoids, will wear the freestyle Libre 2.0 CGM for either 14 consecutive days or their Neuro ICU admission. CGM data will be available in real time to monitor glucose during their hospitalization. Comparison of glucose values from CGM technology and the standard of care fingerstick blood glucose values will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine E Price, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- WakeForest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal